CLINICAL TRIAL: NCT03540667
Title: Prospective Observational Study of Current Perioperative Care for Hip and Knee Arthroplasty in South Africa, and Associated Outcomes
Brief Title: Study of Hip and Knee Arthroplasty in South Africa
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Margot Flint, Medical Researcher, University of Cape Town
Other Study IDs: The BETTER care protocol - 1
Record Dates: First submitted 2018-05-04; First posted 2018-05-30 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip; Arthritis, Rheumatoid; Arthritis Knee; Arthritis of Hip
Keywords: Total hip arthroplasty; Total knee arthroplasty; Total joint arthroplasty; Low middle income country; Enhanced recovery pathway
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group study: The study population will include patients presenting for primary elective unilateral total hip and knee arthroplasty.

SUMMARY:
This multi-site, observational, prospective study aims to investigate current practice and associated outcomes for patients scheduled for elective unilateral total hip or knee arthroplasty in South Africa.This information will provide baseline values, against which effects of implementing a multidisciplinary enhanced care protocol for arthroplasty patients will be compared (the subsequent study).

DETAILED DESCRIPTION:
RESEARCH PROBLEM:

In the past 20 years, enhanced recovery pathways (ERPs) have become increasingly integrated into most surgical fields as standard care in high income countries, as is exemplified by national priority programs and the widespread acceptance of the Enhanced Recovery After Surgery (ERAS) society network. ERPs represent a fundamental shift towards a patient-centred, multidisciplinary-driven continuity of care that aim to attenuate surgical stress and expedite recovery. Studies on total joint arthroplasty (TJA) for both hips and knees have shown that implementation of an evidence-based, structured approach to patient care decreases postoperative morbidity and consequently length of stay without increasing readmission rate.

However, in low- and middle-income countries, the value of implementing ERPs is yet to be explored. This may be because: i) the perception that current hospital resources may make it difficult to develop and implement structured and sustainable protocols to enhance postoperative recovery, and ii) short and long-term data collection on the quality of the work provided is scarce, inhibiting the ability to benchmark clinical results and improve the service provided to patients. Despite these challenges, a healthcare system in a middle-income country such as South Africa may benefit from the implementation of ERPs through reduced postoperative morbidity and the associated cost reductions, as has been demonstrated in high-income countries.

STUDY RATIONAL:

Documentation of current perioperative interventions with associated postoperative outcomes is crucial before implementing a new model for perioperative care. As such, this study will give the investigators baseline values against which the perioperative results achieved from instituting a multidisciplinary enhanced care programme for South African arthroplasty patients will be analyzed.

STUDY DESIGN:

This is a 10-week prospective observational audit of patients scheduled for primary elective unilateral total hip or knee arthroplasty at 9 District, Regional and Central hospitals in South Africa.

PATIENT RECRUITMENT, DATA COLLECTION AND CONFIDENTIALITY:

The patients will be recruited consecutively by the orthopaedic surgeons in the preoperative arthroplasty clinic or when presenting for admission before surgery (minimum 1 day before surgery). Staff from the departments of orthopaedic surgery, physiotherapy and anaesthesia will be responsible for in-hospital data capture. Telephonic follow-up interviews 30 days and 12 months after surgery will be conducted by the Principal Investigator or dedicated research assistants. The patients will be informed that they can choose to leave the study at any time during the study period.

Each individual center will collect and record data on either an electronic or paper case record form (CRF) for every patient recruited. Access to the data entry system will be protected by username and password delivered during the registration process for individual local investigators. All electronic data transfer between participating centres and the coordinating center will be encrypted using a secure protocol (HTTPS/SSL 3.0 or better).

TIME FRAME:

The study will run for 10 weeks at each enrolled site. The in-hospital and 30 day data collection is expected to be completed in 2018.

RISK AND BENEFITS:

Participation in the study will not add any risk to the patient, why the patient's safety is intact. Principles of Helsinki and Good Clinical Practice will be adhered to.

SAMPLE SIZE CALCULATION AND STATISTICAL ANALYSIS:

As knowledge on current postoperative outcomes after hip and knee arthroplasty in South Africa is scarce, this study is a descriptive hypothesis generating study to establish baseline data for future studies, and hence there is no formal power calculation for this study's primary outcome; Days alive and at home 30 days after surgery (DAH30). However, in the study by Myles and colleagues (Myles et al. BMJ Open. 2017; 7(8): e015828. Published online 2017 Aug 18. doi: 10.1136/bmjopen-2017-015828) patient cohorts of approximately 200 patients resulted in clinically relevant and acceptable 95% CI, why we aim to enrol minimum 200 patients. The data are expected to be non-parametric and will be presented as median with interquartile range (25-75 percentile).

As the investigators are unaware of any publications of South African orthopaedic patients which report the specified secondary outcomes, the data will be used to establish a baseline incidence in South African arthroplasty patients for HRQoL (preoperative, 30 days and 12 months postoperative), TUG (in-hospital day 3), mortality (12 months postoperative) and prosthetic joint infection and joint revision (12 months postoperative). These data will be used to power future interventional studies.

Continuous variables will be described using sample mean and standard deviation (SD) and categorical variables using sample median and interquartile range (IQR). Where statistical comparisons are to be made between continuous variables, the unpaired t-test or Mann Whitney U test will be used as appropriate. Categorical data will be compared using the χ2 test.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for primary elective unilateral total hip or knee arthroplasty in the 10 week study period at the 10 participating study sites in South Africa.
* Patients must accept to be contacted telephonically 30 days and 12 months after surgery.

Exclusion Criteria:

* Patients who do not have a mobile telephone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for primary elective unilateral total hip or knee arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
"Days alive and at home 30 days after surgery" (DAH30) | 30 days
  A patient centered measure which integrates length of hospital stay, readmission due to postoperative complications, discharge destination and early death after surgery . This outcome is an overall measure of the recovery profile as it captures much of the surgical experience, integrating efficacy, quality and safety thus reflecting value based care and actions. As such, DAH30 is transparent and can be used for benchmarking performance of quality of perioperative care.

SECONDARY OUTCOMES:
Timed Up and Go test | 2-5 days after surgery
  Timed Up and Go (TUG) is a clinical performance based measure of lower extremity function, mobility and fall risk. It measures how long it takes a patient to get up from a chair, walk 3 meters and return to sitting in the chair. The Physiotherapist will perform TUG on day 3 after surgery. If the patient is discharged earlier, the TUG test will be performed on discharge. If the TUG test can't be performed (ex. lack of personnel on week-ends) the TUG will be performed on day 5 after surgery, unless the patient is discharged earlier than day 5 - in that case the TUG will be performed on discharge.
EQ-5D | 30 days and 1 year after surgery
  Defines health based on 5 dimensions; mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
EQ-VAS | 30 days and 1 year after surgery
  Visual analogue scale (VAS) generates a self-rated Health Related Quality of Life score.
Satisfaction with surgery | 30 days and 1 year after surgery
  To assess overall patient satisfaction with the surgery we will ask the question: "To better understand how satisfied you are with the operation, we would like to know if you would have this operation again, if it were required on the other joint"? (yes/no).
1-year incidence of mortality | 1 year follow up
  Incidence of mortality 1 year after surgery
Prosthetic joint infection rate | 1 year follow up
  Incidence of prosthetic joint infection 1 year after surgery
Joint revision | 1 year follow up
  Incidence of joint revision 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Plenge, MD, Principal Investigator — University of Cape Town
Locations (9):
- South Africa (9):
  - Universitas Academic Hospital, Bloemfontein, Free State
  - Steve Biko Academic Hospital, Pretoria, Gauteng
  - Albert Luthuli Central Hospital, Durban, KwaZulu-Natal
  - Grey's Hospital, Pietermaritzburg, KwaZulu-Natal
  - Mitchells Plain Hospital, Cape Town, Western Cape
  - Somerset Hospital, Cape Town, Western Cape
  - Victoria Hospital, Cape Town, Western Cape
  - Groote Schuur Hospital, Cape Town, Western Cape
  - Paarl Hospital, Paarl, Western Cape

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Plenge U, Parker R, Davids S, Davies GL, Fullerton Z, Gray L, Groenewald P, Isaacs R, Kauta N, Louw FM, Mazibuko A, North DM, Nortje M, Nunes GM, Pebane N, Rajah C, Roos J, Ryan P, September WV, Shanahan H, Siebritz RE, Smit RW, Sombili S, Torborg A, van der Merwe JF, van der Westhuizen N, Biccard B. Quality of recovery after total hip and knee arthroplasty in South Africa: a national prospective observational cohort study. BMC Musculoskelet Disord. 2020 Nov 5;21(1):721. doi: 10.1186/s12891-020-03752-x. PMID 33153453